CLINICAL TRIAL: NCT01432080
Title: Does Increasing Immunosuppression Prevent Transplant-associated Lung-disease Triggered by Viral Respiratory Tract Infection Following Allogeneic Stem Cell Transplant? A Pilot Study
Brief Title: Steroids, Azithromycin, Montelukast, and Symbicort (SAMS) for Viral Respiratory Tract Infection Post Allotransplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not meeting recruitment targets
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: The Canadian Blood and Marrow Transplant Group (Network)
Responsible Party: Principal Investigator, Elizabeth Krakow, Fellow in Hematopoietic Cell Transplantation, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMR1102
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Tract Infections; Bronchiolitis Obliterans; Cryptogenic Organizing Pneumonia; Lung Diseases, Interstitial
Keywords: Pulmonary disease, chronic obstructive; Viral respiratory tract infections; Respiratory syncytial viruses; Influenza virus A; Influenza virus B; Transplantation, Allogeneic
MeSH Terms: conditions — Respiratory Tract Infections; Bronchiolitis Obliterans; Cryptogenic Organizing Pneumonia; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive | interventions — Prednisone; Steroids; Azithromycin; montelukast; Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care includes fluids, antipyretics, ribavirin for RSV infection, and oseltamivir for influenza infection, and intravenous immune globulin for patients with low IgG levels.
- SAMS (Experimental): Subjects randomized to the SAMS arm will receive a four-drug combination (Steroids, Azithromycin, Montelukast, and Symbicort).
  Interventions: Drug: Prednisone; Drug: Azithromycin; Drug: Montelukast; Drug: Symbicort

INTERVENTIONS:
Drug: Prednisone — Prednisone 0.75 mg/kg actual body weight/day PO for 7 days followed by a 7 day taper.
  Other Names: Deltasone; Steroids
  Arms: SAMS
Drug: Azithromycin — Azithromycin 250 mg PO daily for 2 weeks, then 3 times per week until 3 months
  Arms: SAMS
Drug: Montelukast — Montelukast 10 mg PO qhs for 3 months
  Other Names: Singulair
  Arms: SAMS
Drug: Symbicort — Symbicort 200/6 mcg, 2 inhalations every 12 hours for 3 months
  Other Names: Budesonide; Formoterol
  Arms: SAMS

SUMMARY:
For many patients with blood cancers, stem cell transplantation from a family member or from an unrelated donor remains the only potentially curative option. Unfortunately, up to 40% of patients develop chronic lung disease after the transplant, which substantially increases the risk of death in the long-term. Currently, patients with transplant-related lung disease are treated with some combination of steroids and other immunosuppressant drugs, but only about 1 out of 5 improve.

The importance of our study is that the investigators aim to prevent the development of transplant-related chronic lung disease in the first place. Because a strong risk factor for such chronic lung disease is a prior viral respiratory tract infection, the investigators think there is a window of opportunity to intervene. As soon as "cold and flu" symptoms start, the investigators will treat patients with a combination of drugs aimed at eliminating damaging immune responses triggered by the virus. In the absence of such treatment, the investigators believe these lung-damaging immune responses would persist even after the virus disappears. Our hope is that preventive treatment might avoid the development of chronic lung disease, and this would substantially increase long-term survival in our transplant patients.

This is a pilot study. Once feasibility is established, the investigators will seek to expand this study into a definitive clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic transplant within the prior 1 year
* Age greater than or equal to 18 years
* Capable of informed consent
* Neutrophil engraftment has occurred
* This is the first clinically-recognized episode of viral respiratory tract infection after transplant

Exclusion Criteria:

* Proof or high suspicion for bacterial, fungal or any non-viral microorganism causing pneumonia
* CMV, VZV or HSV pneumonia
* Prior diagnosis of a chronic transplant-related non-infectious pulmonary complication (ex: BO, COP)
* Treating physician believes the risk of systemic steroids is too great
* Currently receiving prednisone at or greater than 0.25 mg/kg/day or the equivalent dose of another steroid
* Currently receiving pentostatin
* Mycophenolate initiated de novo or increased within the past 4 weeks
* Use of inhaled corticosteroids within the past 2 weeks for at least 1 week
* Haploidentical or T-cell depleted graft
* Lack of pre-transplant pulmonary function tests
* Evidence of a prior symptomatic viral respiratory tract infection following transplant, whether treated or not
* Allergy or adverse reaction to any of the study drugs
* Relapse or progression of the underlying malignancy
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of new chronic lung disease | 6 months following diagnosis of the viral respiratory tract infection
  The incidence rate of new non-infectious pulmonary complications within the 6 month follow-up period will be calculated. Non-infectious pulmonary complications include new airflow obstruction, new restrictive lung disease, and new mixed obstruction/restriction as measured by spirometry at study enrolment, 2 and 8 weeks following viral infection, and by full pulmonary function tests at 3 and 6 weeks following viral infection.

SECONDARY OUTCOMES:
Prevalence of non-infectious pulmonary complications | 6 months following the diagnosis of viral respiratory tract infection
  Non-infectious pulmonary complications (NIPCs) include airflow obstruction, restrictive lung disease, and mixed obstruction/restriction as determined by pulmonary function tests. The prevalence of NIPCs will be determined among subjects surviving to 6 months post viral respiratory tract infection.
Long-term functional impairment as defined by need for supplemental oxygen | 6 months post viral respiratory tract infection
  The percentage of subjects needing at least 1 month of supplemental oxygen on most days per week, not counting the period of symptomatic viral respiratory tract infection, will be determined in both arms.
Patient-perceived long-term functional impairment | 6 months post viral respiratory tract infection
  A FACT-BMT questionnaire will be administered at baseline and again to subjects surviving 6 months post respiratory tract infection to measure patient-perceived functional impairment.
Time to clearance of viral infection | Every 2 weeks until virus is no longer detectable
  Subjects in whom a respiratory virus is detected will undergo repeat testing every 2 weeks until the virus is no longer detectable. This is an exploratory analysis. The natural history of many of these community-acquired viruses in the transplant population is not known.
Incidence of progression to respiratory failure | 21 days after enrolment
  This endpoint includes admission to hospital because of documented desaturation, need for supplemental oxygen, and need for mechanical ventilation.
Incidence of bacterial or fungal superinfection | Within 21 days after enrolment
  The incidence of secondary bacterial and fungal pneumonias will be compared in the two arms, to verify that the added immunosuppression does not contribute to further infectious complications.
Incidence of various other infectious complications | Within 6 months after enrolment
  The incidence of various other infectious complications, specifically including but not limited to CMV reactivations and CMV disease, zoster, and septicemia will be monitored in both arms.
Overall survival from date of viral respiratory tract infection | 3 months post enrolment
Overall survival from date of viral respiratory tract infection | 6 months post enrolment
Overall survival from date of transplant to end of study follow-up | 6 months post enrolment
Overall survival at 1 year post-transplant | 1 year post-transplant
  This measure will be applied to the group overall and also analyzed according to subgroups of patients presenting viral respiratory tract infections within 30 days of transplant, 31-100 days of transplant, and 101-365 days of transplant.
Cumulative incidence of death attributable to transplant associated lung disease | 6 months post enrolment
Cumulative incidence of death from other causes | 6 months post enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth F Krakow, MD,CM, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital; Sandra Cohen, MD, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital (Hôpital Maisonneuve-Rosemont), Montreal, Quebec, Canada

REFERENCES:
- See also: Maisonneuve-Rosemont Hospital's Stem Cell Transplant Program — http://gmo-hmr.org/en/index.php